CLINICAL TRIAL: NCT01159262
Title: A Phase II/III, Open-Label, Multicenter, Safety, Efficacy and Pharmacokinetic Study of Dexmedetomidine in Neonates Ages ≥28 Weeks to ≤44 Weeks Gestational Age
Brief Title: Safety, Efficacy and Pharmacokinetic Study of Dexmedetomidine in Pediatrics Ages ≥28 Weeks to ≤44 Weeks Gestational Age
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX-09-08
Record Dates: First submitted 2010-06-30; First posted 2010-07-09 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Sedation
Keywords: Initially intubated and mechanically ventilated neonates
MeSH Terms: interventions — Midazolam; Fentanyl; Morphine; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dexmedetomidine 0.05 mcg/kg (Experimental): Dexmedetomidine loading dose 0.05 mcg/kg; maintenance infusion: 0.05 mcg/kg/hr.
  Interventions: Drug: Midazolam; Drug: Fentanyl/Morphine; Drug: Dexmedetomidine
- Dexmedetomidine 0.1 mcg/kg (Experimental): Dexmedetomidine loading dose: 0.1 mcg/kg; maintenance infusion 0.1 mcg/kg/hr.
  Interventions: Drug: Midazolam; Drug: Fentanyl/Morphine; Drug: Dexmedetomidine
- Dexmedetomidine 0.2 mcg/kg (Experimental): Dexmedetomidine loading dose 0.2 mcg/kg; maintenance infusion 0.2 mcg/kg/hr.
  Interventions: Drug: Midazolam; Drug: Fentanyl/Morphine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — Per package insert, N-PASS (Neonatal Pain, Agitation, and Sedation Scale) scores and investigator discretion
Drug: Fentanyl/Morphine — Per package insert, N-PASS scores and investigator discretion.
Drug: Dexmedetomidine
  Other Names: Precedex

SUMMARY:
The purpose of this study is to investigate the safety, efficacy and pharmacokinetics (PK) of dexmedetomidine (DEX) at 3 different dose levels in infants, ages ≥28 weeks to ≤44 weeks gestational age, administered as a loading dose followed by a continuous infusion for a minimum of 6 hours and up to 24 hours in the neonatal intensive care unit (NICU), cardiac intensive care unit (CICU), or pediatric intensive care unit (PICU).

ELIGIBILITY:
Inclusion Criteria:

1. Initially intubated and mechanically ventilated pediatric subjects in an intensive care setting anticipated to require a minimum of 6 hours of continuous IV sedation.
2. The ability to complete all PK sampling blood draws.
3. Age: subjects must fit into 1 of the following age ranges at screening:

   * Preterm neonates ≥28 weeks through <36 weeks, gestational age; this would constitute treatment Group I.
   * Term neonates born at ≥36 weeks through ≤44 weeks gestational age; this would constitute treatment Group II.
4. Weight: subject's weight at the time of enrollment must be >1000 g.
5. Subject's parent(s) or legal guardian(s) has/have voluntarily signed and dated the informed consent document approved by the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).

Exclusion Criteria:

1. Neonate subjects with neurological conditions that prohibit an evaluation of sedation such as:

   * Diminished consciousness from increased intracranial pressure.
   * The presence of catastrophic brain injury or other severe mental disorders that would make responses to sedatives unpredictable and/or measurement of the N-PASS unreliable.
   * Subjects with immobility from neuromuscular disease or continuous infusion of neuromuscular blocking (NMB) agents.
2. Subjects with second degree or third degree heart block unless subject has a pacemaker or pacing wires are in situ.
3. Heart rate <120 bpm prior to the initiation of study drug.
4. Exposure to any investigational drug within 30 days prior to study drug administration.
5. Previous exposure to Dexmedetomidine (DEX) as part of an investigational study.
6. Maternal history of poly-substance drug abuse, based upon the presence of 1) an abnormal urine drug screen for cocaine, opiates and/or benzodiazepines; or 2) Investigator's judgment.
7. At the discretion of the Investigator, subjects in whom the risk of DEX treatment is expected to exceed its benefits.
8. Subjects who have a known allergy or contraindication to fentanyl, morphine, Midazolam, DEX, or other α-2 agonists.
9. Requirement for medications other than DEX, Midazolam, morphine, or fentanyl for sedation and pain control.
10. Screening alanine aminotransferase (ALT) levels >115 U/L.

Ages: 28 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (17):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - University of California San Francisco, Department of Pediatrics, Division of Neonatology, San Francisco, California
  - Dept. of Anesthesia, SUMC, Stanford, California
  - University of Miami - Miller School of Medicine, Department of Anesthesiology, Miami, Florida
  - Georgia Health Sciences University, Augusta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Loyola University Medical Center, Maywood, Illinois
  - Wichita, Kansas
  - Kosair Charities Pediatric Clinical Research Unit, University of Louisville, Louisville, Kentucky
  - Duke University Medical Center, Department of Anesthesiology, Durham, North Carolina
  - Akron Children's Hospital Medical Center, Akron, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Greenville, South Carolina
  - West Virginia University School of Medicine, Morgantown, West Virginia
- Zona 11 Guatemala, Guatemala

REFERENCES:
- [Derived] Chrysostomou C, Schulman SR, Herrera Castellanos M, Cofer BE, Mitra S, da Rocha MG, Wisemandle WA, Gramlich L. A phase II/III, multicenter, safety, efficacy, and pharmacokinetic study of dexmedetomidine in preterm and term neonates. J Pediatr. 2014 Feb;164(2):276-82.e1-3. doi: 10.1016/j.jpeds.2013.10.002. Epub 2013 Nov 14. PMID 24238862

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine 0.05 mcg/kg: Dexmedetomidine loading dose 0.05 mcg/kg; maintenance infusion: 0.05 mcg/kg/hr.
  Midazolam: Per package insert, N-PASS (Neonatal Pain, Agitation, and Sedation Scale) scores and investigator discretion
  Fentanyl: Per package insert, N-PASS scores and investigator discretion.
  Dexmedetomidine
- Dexmedetomidine 0.1 mcg/kg: Dexmedetomidine loading dose: 0.1 mcg/kg; maintenance infusion 0.1 mcg/kg/hr.
  Midazolam: Per package insert, N-PASS scores and investigator discretion
  Fentanyl: Per package insert, N-PASS scores and investigator discretion.
  Dexmedetomidine
- Dexmedetomidine 0.2 mcg/kg: Dexmedetomidine loading dose 0.2 mcg/kg; maintenance infusion 0.2 mcg/kg/hr.
  Midazolam: Per package insert, N-PASS scores and investigator discretion
  Fentanyl: Per package insert, N-PASS scores and investigator discretion.
  Dexmedetomidine
Period: Overall Study
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Started | 14 | 14 | 8
Completed | 14 | 14 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dexmedetomidine 0.05 mcg/kg: Dexmedetomidine loading dose 0.05 mcg/kg; maintenance infusion: 0.05 mcg/kg/hr.
  Midazolam: Per package insert, N-PASS scores and investigator discretion
  Fentanyl: Per package insert, N-PASS scores and investigator discretion.
  Dexmedetomidine
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg | Total
Number analyzed (Participants) | 14 | 14 | 8 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 8 | 36
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 1.637 (1.8290) | 1.098 (1.0849) | 2.225 (1.5779) | 1.558 (1.5382)
Age, Customized [Number; unit: Participants]
  = 28 weeks to < 36 weeks gestational age | 6 | 6 | 0 | 12
  >= 36 weeks to <= 44 weeks gestational age | 8 | 8 | 8 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 0 | 12
  Male | 8 | 8 | 8 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 10 | 10 | 6 | 26
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 3 | 3 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Received Rescue Medication Midazolam for Sedation During Dexmedetomidine Infusion
Time Frame: During study drug administration (6 to 24 hours)
Population: Efficacy Evaluable Population: All subjects who received randomized Dexmedetomidine for at least 6 hours.
Measure: Number; unit: percentage of subjects
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Number analyzed (Participants) | 14 | 14 | 8
percentage of subjects | 7.1 | 7.1 | 25

2. Secondary Outcome: Percentage of Subjects Who Received Rescue Medication for Analgesia During Dexmedetomidine Infusion
Time Frame: During Study drug administration (6 to 24 hours)
Population: Efficacy Evaluable Population: All subjects who received randomized Dexmedetomidine for at least 6 hours.
Measure: Number; unit: percentage of subjects
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Number analyzed (Participants) | 14 | 14 | 8
percentage of subjects | 35.7 | 35.7 | 75

3. Secondary Outcome: Total Amount of Rescue Medication Midazolam Given for Sedation During Dexmedetomidine Infusion (Among Who Used)
Time Frame: During Study drug administration (6 to 24 hours)
Population: All subjects who received midazolam during Dexmedetomidine infusion
Measure: Mean (Standard Deviation); unit: Milligram
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Number analyzed (Participants) | 1 | 1 | 2
Milligram | .360 (NA) — Only 1 subject received rescue medication in the group. Standard deviation is not able to be calculated. | .500 (NA) — Only 1 subject received rescue medication in the group. Standard deviation is not able to be calculated | 1.125 (1.4637)

4. Secondary Outcome: Total Amount of Rescue Medication Fentanyl Given for Sedation During Dexmedetomidine Infusion (Among Who Used)
Time Frame: During study drug administration (6 to 24 hours)
Population: All subjects who received fentanyl during Dexmedetomidine infusion
Measure: Mean (Standard Deviation); unit: Microgram
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Number analyzed (Participants) | 5 | 3 | 5
Microgram | 10.808 (7.1305) | 5.667 (3.5119) | 9.522 (7.5131)

5. Secondary Outcome: Total Amount of Rescue Medication Morphine Given for Sedation During Dexmedetomidine Infusion (Among Who Used)
Time Frame: During study drug administration (6 to 24 hours)
Population: All subjects who received morphine during Dexmedetomidine infusion
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Number analyzed (Participants) | 0 | 2 | 3
milligram |  | 0.275 (0.0354) | 0.400 (0.1732)

6. Secondary Outcome: Weight-adjusted Total Amount (Per kg) of Rescue Medication Midazolam Given for Sedation During Dexmedetomidine Infusion (Among Who Used)
Time Frame: During study drug administration (6 to 24 hours)
Population: All subjects who received midazolam during Dexmedetomidine infusion
Measure: Mean (Standard Deviation); unit: milligrams/Kg
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Number analyzed (Participants) | 1 | 1 | 2
milligrams/Kg | 0.100 (NA) — Only 1 subject received rescue medication in the group. Standard Deviation was not able to be calculated | 0.152 (NA) — Only 1 subject received rescue medication in the group. Standard Deviation was not able to be calculated | 0.318 (0.4133)

7. Secondary Outcome: Weight-adjusted Total Amount (Per kg) of Rescue Medication Fentanyl Given for Analgesia During Dexmedetomidine Infusion (Among Who Used)
Time Frame: During study drug administration (6 to 24 hours)
Population: All subjects who received fentanyl during Dexmedetomidine infusion
Measure: Mean (Standard Deviation); unit: microgram/Kg
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Number analyzed (Participants) | 5 | 3 | 5
microgram/Kg | 5.137 (6.3696) | 1.863 (0.8761) | 2.725 (2.1383)

8. Secondary Outcome: Weight-adjusted Total Amount (Per kg) of Rescue Medication Morphine Given for Analgesia During Dexmedetomidine Infusion (Among Who Used)
Time Frame: During study drug administration (6 to 24 hours)
Population: All subjects who received morphine during Dexmedetomidine infusion
Measure: Mean (Standard Deviation); unit: milligram/Kg
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Number analyzed (Participants) | 0 | 2 | 3
milligram/Kg |  | 0.125 (0.0348) | 0.109 (0.0540)

9. Secondary Outcome: Time to Successful Extubation in DEX-exposed Subjects
Time Frame: From start of DEX administration to extubation of each subject up to 7 days post-infusion
Population: Efficacy Evaluable Population: All subjects who received randomized Dexmedetomidine for at least 6 hours.
Measure: Median (95% Confidence Interval); unit: hour
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Number analyzed (Participants) | 14 | 14 | 8
hour | 22.9 [4.467 to 100.67] | 49.3 [33.167 to 79.583] | 23.7 [4.667 to 67.333]

ADVERSE EVENTS:
Time Frame: Start of study drug administration until 7 days following the start of study drug. Serious adverse events collected from signing of informed consent until 7 days following start of study drug administration or hospital discharge (whichever comes first).
Description: Patients were monitored for safety parameters from 6 to 24 hours in the ICU.
Arm/Group | Dexmedetomidine 0.05 mcg/kg | Dexmedetomidine 0.1 mcg/kg | Dexmedetomidine 0.2 mcg/kg
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/14 | 0/8
Other Adverse Events (participants affected / at risk) | 7/14 | 9/14 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine 0.05 mcg/kg (N=14) | Dexmedetomidine 0.1 mcg/kg (N=14) | Dexmedetomidine 0.2 mcg/kg (N=8)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.8% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine 0.05 mcg/kg (N=14) | Dexmedetomidine 0.1 mcg/kg (N=14) | Dexmedetomidine 0.2 mcg/kg (N=8)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbiliruninaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Shunt stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Hemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 3 (3) | 3 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Plueral effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diastolic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No